CLINICAL TRIAL: NCT03949595
Title: Rapid Eating Is Linked to Emotional Eating in Obese Women Relieving From Bariatric Surgery
Acronym: BS-Women
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2018Ao004
Record Dates: First submitted 2019-05-13; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Obesity
Keywords: Obese; Food behaviour; Eating rate
MeSH Terms: conditions — Obesity | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cases: women suffering from severe/massive obesity
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection

SUMMARY:
The aim of the study was to analyse eating rate in comparison to other aspects of eating habits in women suffering from severe/massive obesity.

DETAILED DESCRIPTION:
Eating rate is associated with BMI and weight gain in various populations and is a factor modulating the risk of complications after bariatric surgery. The aim of the present study is to determine whether common difficulties to change eating rate in subjects with obesity candidate to bariatric surgery could be due to more extensive abnormalities in eating behaviour.

ELIGIBILITY:
inclusion criteria :

* BMI ≥ 35 kg/m
* responses to a self-administered questionnaire distributed between November 2011 and March 2014 to female patients attending a nutrition consultation for overweight, or attending an outpatient visit prior to bariatric surgery, both within the Champagne-Ardenne Specialized Obesity Clinic, at the University Hospital Robert Debré in Reims, France
* Patients who agree to participate to the study
* Major patient

exclusion criteria :

* Patient under law protection
* Minor patient
* Patients with uncontrolled diabetes (HbA1c ≥ 8.0% at inclusion) or those treated with glucagon-like peptide-1 (GLP-1) receptor antagonists, as well as patients treated by glucocorticoids (their current treatment was systematically reported)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women suffering from obesity and their eating habits
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2014-03-01 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
Eating Rate | Day 0
  Eating Rate was assessed by using an analog scale from 1 (slowest eating) to 10 (fastest eating)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Canterini CC, Gaubil-Kaladjian I, Vatin S, Viard A, Wolak-Thierry A, Bertin E. Rapid Eating is Linked to Emotional Eating in Obese Women Relieving from Bariatric Surgery. Obes Surg. 2018 Feb;28(2):526-531. doi: 10.1007/s11695-017-2890-4. PMID 28871527